CLINICAL TRIAL: NCT00434876
Title: The Effects of Quetiapine on Sleep During Alcohol Abstinence
Brief Title: The Effects of Quetiapine (Seroquel XR) on Sleep During Alcohol Abstinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Subhajit Chakravorty (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Subhajit Chakravorty, Staff Physician, Corporal Michael J. Crescenz VA Medical Center
Organization: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101206
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-07

CONDITIONS: Alcoholism; Sleep Initiation and Maintenance Disorders
Keywords: Alcoholism; Insomnia; Quetiapine; Seroquel
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine XR
  Interventions: Drug: Quetiapine XR
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo.

INTERVENTIONS:
Drug: Quetiapine XR — Quetiapine is a second generation antipsychotic medication, which has also recently shown to be associated with properties of mood stabilization in bipolar disorder.
  Other Names: Seroquel XR
  Arms: 1
Drug: Placebo. — Inactive or inert pill which will be used as a comparator.
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine how efficacy of quetiapine (seroquel XR) in improving the sleep in recovering alcohol dependent subjects.

DETAILED DESCRIPTION:
Sober alcohol dependent subjects frequently complain of difficulty falling asleep as well as staying asleep which may eventually lead to relapse. Novel antipsychotic medications such as quetiapine have shown some efficacy in treating alcoholism and have also shown some benefit in improving insomnia.

The primary aim of this study is to determine the degree to which quetiapine improves sleep in veterans during the early phase of recovery from alcohol dependence. The sleep efficiency from an in-lab polysomnogram will be the primary outcome measure. Secondary measures of sleep will include the Pittsburgh Sleep Quality Index, Insomnia Severity Index, and actigraphy. Other additional aims will explore for alcohol use and cravings, change in psychiatric symptoms using the The Time Line Follow Back measure, Penn Alcohol Craving Scale (PACS), the Patient Health Questionnaire-9 item scale (PHQ-9), and the Beck's Anxiety Inventory (BAI) respectively.

Twenty four subjects within the first year of sobriety will be enrolled. Participants will be undergo an extensive baseline screening procedure. After 2 consecutive in-laboratory polysomnograms they will be treated with either Quetiapine XR or matching placebo pills targetting a dose of 400 mg a night. The treatment duration will be 8 weeks and during the eight week of treatment they will undergo 2 more nights of in-laboratory polysomnogram. All subjects will also receive Medical Management therapy, a standardized psychosocial intervention which is medically-based and focusses on alcohol abstinence and medication compliance.

ELIGIBILITY:
Inclusion Criteria: subjects between the ages of 18-65 years, with a DSM-IV diagnosis of current alcohol dependence (past year), can speak, understand, and print in English, and is capable of giving written informed consent

Exclusion Criteria: Positive urine drug screen for opioids, cocaine, or amphetamine (excluding THC), dependence on other drugs excluding alcohol/nicotine/cannabis over the past year, unstable psychiatric, medical disorders, cataracts [posterior capsular/ nuclear (grade NS3 or more), currently on any maintenance psychotropic medications affecting sleep, currently pregnant, nursing, or not using a reliable method of contraception; history of hypersensitivity to antipsychotic drugs, including quetiapine, severe cognitive impairment, severe untreated obstructive sleep apnea, and inadequately controlled diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhajit Chakravorty, MD, Principal Investigator — Philadelphia, OPC
Locations (1):
- Philadelphia, OPC, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Addiction psychiatry clinic, behavioral health laboratory, and self referrals solicited through flyers.
Groups:
- Quetiapine XR: The pills were taken at bedtime and the dose was titrated flexibly in the following fashion over the first week: 50 mg dose for 2 nights, followed by 200 mg a night for 2 nights, and then 300 mg a night for 2 nights and to a final dose of 400 mg daily starting on night # 7. Medication taper commenced at week 8 in the reverse stepwise fashion after the second set of two polysomnograms.
- Placebo: The matching placebo pills were similarly taken at bedtime and the dose was titrated flexibly in the following fashion over the first week: 50 mg dose for 2 nights, followed by 200 mg a night for 2 nights, and then 300 mg a night for 2 nights and to a final dose of 400 mg daily starting on night # 7. Medication taper commenced at week 8 in the reverse stepwise fashion after the second set of two polysomnograms.
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine: Quetiapine XR
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (6) | 51 (8) | 52 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency (From an In-laboratory Polysomnogram)
Description: The fraction of time spent asleep to the total time in bed (%).
Time Frame: Baseline, and week 8 of treatment.
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Quetiapine XR: Quetiapine XR
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 10 | 10
percentage
  Sleep Efficiency (baseline) | 70.70 (17.49) | 78.63 (12.89)
  Sleep Efficiency (after 8 weeks of treatment) | 79.45 (16.52) | 82.80 (11.57)
Statistical Analysis 1: Comparison: Quetiapine XR vs Placebo; Test type: Superiority or Other; p = 0.49, Mixed Models Analysis

2. Secondary Outcome: Insomnia Severity Index (ISI)
Description: ISI total score; this scale assesses for global insomnia severity (range 0-24). Higher scale scores indicate higher insomnia severity.
Time Frame: Baseline, weeks 1, 3, 5, and 7 of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  ISI (baseline) | 17.00 (4.08) | 14.80 (7.14)
  ISI (week 7) | 5.40 (4.83) | 6.70 (7.34)
Statistical Analysis 1: Comparison: Quetiapine XR vs Placebo; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: PSQI total score (range 0-21). A PSQI total score > 5 indicates insomnia, with higher scores denoting a decrease in sleep quality.
  The PSQI global score assesses for the overall quality of sleep and is computed by adding the 7 component scale scores. This widely used 19-item self-rated scale evaluates the subjective quality of sleep over the last 4 weeks. The PSQI was administered at baseline, and weeks 4, and 9.
Time Frame: Baseline, weeks 4, and 9.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  PSQI (baseline) | 14.70 (1.94) | 14.60 (1.71)
  PSQI (week 4) | 13.20 (2.61) | 13.80 (2.04)
  PSQI (week 9) | 14.50 (2.56) | 13.80 (2.78)
Statistical Analysis 1: Comparison: Quetiapine XR vs Placebo; Test type: Superiority or Other; p = 0.57, Mixed Models Analysis

4. Secondary Outcome: Wake After Sleep Onset Time (WASO) From an In-laboratory Polysomnogram.
Description: The amount of time spent awake after initially falling asleep and before final awakening (in minutes). None to a fewer minutes is better (than a higher number of minutes).
Time Frame: Baseline, and week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 10 | 10
minutes
  WASO (baseline) | 101.87 (81.80) | 61.17 (37.77)
  WASO (week 8) | 60.71 (71.41) | 66.99 (60.62)
Statistical Analysis 1: Comparison: Quetiapine XR vs Placebo; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Quetiapine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/10
Other Adverse Events (participants affected / at risk) | 7/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=10) | Placebo (N=10)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Relapse to heavy alcohol use leading to inpatient admission (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine (N=10) | Placebo (N=10)
Somnolence (Psychiatric disorders) | 7 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Increased apetite (Psychiatric disorders) | 1 | 0
Dizziness (Cardiac disorders) | 1 | 1
Somatic pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Decreased motivation (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The limitations of this study include the small sample size, and assessment of PSQI, PHQ-9, BAI, and SF-12 at week 9 (immediately after washout from the study drug). The corruption of stored online actigraphic sleep data prevented its interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No